CLINICAL TRIAL: NCT00346658
Title: Magnesium Supplementation to Prevent Bone Loss
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RR16047; 5K23RR016047 (NIH)
Record Dates: First submitted 2006-06-28; First posted 2006-06-30 (Estimated); Last update posted 2008-12-15 (Estimated); Status verified 2008-12

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; bone density; magnesium; vitamin D
MeSH Terms: conditions — Osteoporosis | interventions — Magnesium

INTERVENTIONS:
Drug: magnesium

SUMMARY:
Extreme magnesium deficiency is known to have an impact on the synthesis, secretion and/or action of calcium regulating hormones. Many older adults are at risk for less severe magnesium deficiency, since the majority of adults receive less than the Recommended Daily Allowance of magnesium. We hypothesize that magnesium supplementation will have a beneficial effect on calcium regulating hormones and markers of bone turnover.

DETAILED DESCRIPTION:
This is a 12 month randomized, double-blind, placebo-controlled study of magnesium supplementation. Our hypothesis was that magnesium supplementation would decrease bone turnover markers and alter calcium-regulating hormones: parathyroid hormone and 1, 25 dihydroxyvitamin D.

Male and female adults over 55 without with a T-score at the hip above -2 are randomized to magnesium 250 mg BID or identical placebo BID. At baseline, all participants had a bone mineral density (BMD) by DXA scan at the hip and spine, blood biomarkers of bone resorption and formation, and calcium regulating hormones. Participants were followed for 12 months, with repeat measurement of calcium regulating hormones and bone turnover markers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy ambulatory men and women between the ages of 55-75 years
2. Women at least 5 years after menopause

Exclusion Criteria:

1. Inability to give informed consent in accordance with institutional guidelines
2. Creatinine greater than or equal to 2 mg/dl, since magnesium is excreted by the kidneys
3. Diarrhea or loose frequent stools (> 2 a day) at least 3 days/ week in last 3 months
4. Use within 12 months of estrogen, bisphosphonates, calcitonin, or raloxifene
5. Current use of loop diuretics
6. Use within 12 months of corticosteroids
7. History of hyperparathyroidism, hyperthyroidism, or osteomalacia within past 12 month
8. Vitamin D deficient as measured by 25-hydroxyvitamin D outside of the normal range
9. Magnesium supplementation of greater than 250 mg/day
10. Calcium supplementation of greater than 1500 mg/day
11. Conditions which, in the opinion of the investigator, would interfere with the evaluation of BMD at the spine including severe scoliosis, osteophytosis and lumbar fusion
12. Bilateral hip replacement
13. BMD at the lumbar spine L2-L4 of less than 0.859g/cm2 for women or 0.895 g/cm2 in men; or total hip less than 0.698 g/cm2 for women or 0.731 g/cm2 for men; or femoral neck less than 0.627 g/cm2 for women or 0.658 g/cm2 for men This represents a T-score of less than -2 at each site
14. High serum calcium on screening blood test

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74
Dates: Start 2002-07; Study Completion 2006-09

PRIMARY OUTCOMES:
Biomarkers bone turnover (P1NP and CTX)
Calcium regulating hormones (PTH and 1,25 dihydroxyvitamin D)

SECONDARY OUTCOMES:
Change in BMD at the spine, femoral neck and total hip by DXA
Change in RBC magnesium

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn M Ryder, MD, MS, Principal Investigator — University of Tennessee Health Sciences Center
Locations (1):
- University of Tennessee Health Sciences Center, Memphis, Tennessee, United States